CLINICAL TRIAL: NCT03954002
Title: Quantification of Right Ventricular Function Using Simultaneous Transthoracic and Transoesophageal Echocardiography
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Principal Investigator left
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2018/00987
Record Dates: First submitted 2019-04-29; First posted 2019-05-17 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2021-10

CONDITIONS: Cardiac Surgery
Keywords: Transthoracic Echocardiography (TTE); Transoesophageal Echocardiography (TOE)
MeSH Terms: interventions — Echocardiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TTE and TOE (Experimental): A small flexible tube (TOE probe) will be inserted into your oesophagus, or food pipe, to take images of your heart as per routine anaesthetic care for cardiac surgery.
  Just before and after general anaesthesia is administered, a short transthoracic echocardiography (TTE scan will be performed to acquire images of your heart. This is an ultrasound scan of your heart using a probe on the outside of the chest. During this period, relevant haemodynamic data such as blood pressure and heart rate will be recorded.
  Interventions: Diagnostic Test: TTE and TOE

INTERVENTIONS:
Diagnostic Test: TTE and TOE — A small flexible tube (TOE probe) will be inserted into your oesophagus, or food pipe, to take images of your heart as per routine anaesthetic care for cardiac surgery.
  Just before and after general anaesthesia is administered, a short transthoracic echocardiography (TTE scan will be performed to acquire images of your heart. This is an ultrasound scan of your heart using a probe on the outside of the chest. During this period, relevant haemodynamic data such as blood pressure and heart rate will be recorded.

SUMMARY:
The aims of this study are to evaluate the usefulness of various methods of quantifying right ventricular (RV) function using perioperative transoesophageal echocardiographic (TOE), compared with simultaneous transthoracic echocardiographic (TTE) findings.

DETAILED DESCRIPTION:
The hypothesis of this study that perioperative TOE is useful in quantifying RV function, and that the quantification methods used will correlate well to commonly used, well-studied TTE parameters obtained simultaneously, under the same loading conditions.

Assessment of RV function is of particular importance in the perioperative period. RV dysfunction can be due to a myriad of causes - myocardial ischemia, pulmonary embolism, pulmonary hypertension, congenital heart disease, or cardiomyopathy. The presence of RV failure can lead to difficulty in separation from cardiopulmonary bypass in cardiac surgical patients, and has been shown to be an independent predictor of mortality in high-risk cardiac surgery patients. Additionally, correct identification of RV dysfunction is crucial in order for the correct treatment to be administered. RV failure can lead to underfilling of the left ventricle, and mimic hypovolaemia with hypotension and an exaggerated stroke volume variation. In such a case, failure to diagnose RV dysfunction can wrongly lead to fluid loading and further worsening of right ventricular failure.

While evaluation of right heart function is well described in TTE studies, there is insufficient data at present to recommend a reliable method to quantify RV function using TTE.

In addition to traditional measurements of RV function, we hope to study the usefulness of speckle tracking and strain imaging in assessment of RV function, modalities of echocardiographic image analysis which have garnered increasing interest in recent years.

ELIGIBILITY:
Inclusion Criteria:

* Age > 21 years
* Undergoing elective cardiac surgery
* Planned for intraoperative TOE

Exclusion Criteria:

* Patient refusal
* Emergency surgery
* Haemodynamic instability
* Previous tricuspid valve surgery
* Severe tricuspid regurgitation
* Rhythm other than sinus
* Previous oesophageal / gastric surgery
* Oesophageal stricture / tumour
* Oesophageal diverticulum / fistula
* Active upper GI haemorrhage
* Oesophageal varices

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Data collection of views obtained from TTE | Intra-operatively during general anaesthesia
  Evaluate the usefulness of various methods of quantifying right ventricular (RV) function using perioperative transoesophageal echocardiographic (TOE), compared with simultaneous transthoracic echocardiographic (TTE) findings.
  The main data to be collected for TTE are:
  Pre-induction A4Ch (4 beats), Pre-induction M-mode (lateral TA), Post-induction A4Ch (4 beats), Post-induction M-mode (lateral TA), Post-induction TDI (lateral TA) (PWD)
Data collection of views obtained from TOE | Intra-operatively during general anaesthesia
  Evaluate the usefulness of various methods of quantifying right ventricular (RV) function using perioperative transoesophageal echocardiographic (TOE), compared with simultaneous transthoracic echocardiographic (TTE) findings.
  The main data to be collected for TOE are:
  RV focused ME4Ch (4 beats), M-mode (ME4Ch, lateral TA), TDI (ME4Ch, lateral TA) (PWD), Deep TG RV apical view (4 beats), M-mode (DTG, lateral TA), TDI (DTG, lateral TA) (PWD)

CONTACTS AND LOCATIONS:
Overall Officials: Chang Chuan Melvin Lee, MBBS, MMed, Principal Investigator — National University Health System
Locations (1):
- National University Health System, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Flo Forner A, Hasheminejad E, Sabate S, Ackermann MA, Turton EW, Ender J. Agreement of tricuspid annular systolic excursion measurement between transthoracic and transesophageal echocardiography in the perioperative setting. Int J Cardiovasc Imaging. 2017 Sep;33(9):1385-1394. doi: 10.1007/s10554-017-1128-9. Epub 2017 Apr 13. PMID 28409259
- [Background] Korshin A, Gronlykke L, Nilsson JC, Moller-Sorensen H, Ihlemann N, Kjoller M, Damgaard S, Lehnert P, Hassager C, Kjaergaard J, Ravn HB. The feasibility of tricuspid annular plane systolic excursion performed by transesophageal echocardiography throughout heart surgery and its interchangeability with transthoracic echocardiography. Int J Cardiovasc Imaging. 2018 Jul;34(7):1017-1028. doi: 10.1007/s10554-018-1306-4. Epub 2018 Jan 30. PMID 29383465
- [Background] Tousignant C, Kim H, Papa F, Mazer CD. Evaluation of TAPSE as a measure of right ventricular output. Can J Anaesth. 2012 Apr;59(4):376-83. doi: 10.1007/s12630-011-9659-3. PMID 22302303
- [Background] Bartels K, Karhausen J, Sullivan BL, Mackensen GB. Update on perioperative right heart assessment using transesophageal echocardiography. Semin Cardiothorac Vasc Anesth. 2014 Dec;18(4):341-51. doi: 10.1177/1089253214522326. Epub 2014 Feb 13. PMID 24525287
- [Background] Kasper J, Bolliger D, Skarvan K, Buser P, Filipovic M, Seeberger MD. Additional cross-sectional transesophageal echocardiography views improve perioperative right heart assessment. Anesthesiology. 2012 Oct;117(4):726-34. doi: 10.1097/ALN.0b013e318269054b. PMID 22902962
- [Background] Horton KD, Meece RW, Hill JC. Assessment of the right ventricle by echocardiography: a primer for cardiac sonographers. J Am Soc Echocardiogr. 2009 Jul;22(7):776-92; quiz 861-2. doi: 10.1016/j.echo.2009.04.027. PMID 19560657
- [Background] Forner FA, Hasheminejad E, Dobrovie M, Da Rocha e Silva J, Ender J. Agreement of tricuspid annular systolic excursion (TAPSE) measurement in m-mode between transthoracic (TTE) and transoesophageal (TOE) echocardiography. J Cardiothorac Vasc Anesth 2015; 29 (S2):S31-S58 OP-005